CLINICAL TRIAL: NCT07038850
Title: Improving Caregivers' Adherence to a Sedation-analgesia Protocol Managed by Pediatric Intensive Care Nurses: a Quality Approach Program
Brief Title: Improving Adherence to the Sedation-analgesia Protocol in Pediatric Intensive Care
Acronym: SEDATIDE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL18_0108
Record Dates: First submitted 2025-05-20; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-05

CONDITIONS: Mechanical Ventilation; Analgesia; Nurse Training
Keywords: Nurse driven sedation-analgesia protocols; Adherence to protocol; Pediatric intensive care
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Multimodal nurse training about nurse driven sedation-analgesia protocol — The training program for nursing staff in the use of the sedation-analgesia protocol includes 3 stages:
  1. Initial training: e-learning module to be validated
  2. Feedback session: sessions in small groups of 5 to 6 participants, led by a nurse trainer, allowing interprofessional transmission (questions/answers and critical analyzes of sedation collection sheets).
  3. Bedside rehearsal: individual practice of the sedation-analgesia protocol at the patient's bedside under the supervision of a doctor or nurse trainer.

SUMMARY:
Sedation-analgesia is a major concern in the management of children in pediatric intensive care units (PICUs). International guidelines recommend the use of sedation-analgesia protocols, as their implementation has already proven effective in pediatrics. However, maintaining their long-term application remains a challenge. Indeed, healthcare teams adherence to these protocols tends to decrease over time, thereby compromising their long-term impact. This study aims to evaluate the impact of multimodal nurses training on improving and sustaining adherence to sedation-analgesia protocols. This is a non-randomized, before-and-after interventional prospective study conducted in two mixed pediatric intensive care units (Lyon and Nantes). The investigators seek to evaluate sedation practices before and after the implementation of specific multimodal training for nurses on the sedation-analgesia protocol. The primary outcome is protocol adherence. Secondary outcomes include the duration of mechanical ventilation and PICU stay, the number of daily COMFORT-B score assessments, total medication doses, the incidence of ventilator-associated pneumonia, and a qualitative analysis of non-adherence factors.

ELIGIBILITY:
Inclusion Criteria :

* patients aged 0 to 18 years
* admitted to the PICU
* requiring mechanical ventilation
* receiving continuous sedation for more than 24 hour

Exclusion Criteria :

* patients requiring mechanical ventilation for more than 15 days
* transferred from another unit where sedation had already been initiated
* patients under sedation as part of withdrawing and withholding life-sustaining treatment
* deceased patients
* preexisting tracheostomies

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 285 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Protocol adherence before and after nurse training: daily percentage of therapeutic adjustments in compliance with the sedation-analgesia protocol. | Compliance of therapeutic adjustments with the sedation-analgesia protocol is evaluated over the entire duration of mechanical ventilation. Daily , from initiation of mechanical ventilation until extubation
  Sedation management is considered adequate (when dose increases, decreases, or maintenance are appropriate based on the COMFORT-B score), and inadequate (when adjustments are inappropriate or if the COMFORT-B score is not recorded despite a prescribed target). Cases where no target score is prescribed are excluded from the adherence analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Fabienne BORDET Dr Fabienne BORDET, Doctor, Principal Investigator — HCL
Locations (2):
- France (2):
  - Service de réanimation pédiatrique du CHU de Lyon, Lyon
  - Service de réanimation pédiatrique du CHU de Nantes, Nantes